CLINICAL TRIAL: NCT06804356
Title: Long-term Outcome of Partial Trapeziectomy With Interposition of Poly-L/D-lactide Scaffold (RegJoint) vs. Autologous Tendon for Inflammatory Trapeziometacarpal Joint Arthritis.
Brief Title: Poly-L/D-lactide Implant (RegJoint) Versus Tendon Interposition for Trapeziometacarpal Inflammatory Arthritis: a 15-year Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Thomas Mikael Hackenberg, Doctoral student, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/575/2019
Record Dates: First submitted 2025-01-07; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tendon interposition arthroplasty (Active Comparator): Trapeziometacarpal arthroplasty using autologous tendon interposition to fill the space left by resecting affected joint surfaces.
  Interventions: Procedure: Tendon interposition arthroplasty
- Poly-L-D-lactic acid implant (RegJoint) interposition arthroplasty (Active Comparator): Trapeziometacarpal arthroplasty using poly-L-D-lactic acid implant (RegJoint) interposition to fill the space left by resecting affected joint surfaces.
  Interventions: Procedure: Poly-L-D-lactic acid implant (RegJoint) interposition arthroplasty

INTERVENTIONS:
Procedure: Tendon interposition arthroplasty — Trapeziometacarpal arthroplasty using autologous tendon interposition to fill the space left by resecting affected joint surfaces.
  Arms: Tendon interposition arthroplasty
Procedure: Poly-L-D-lactic acid implant (RegJoint) interposition arthroplasty — Trapeziometacarpal arthroplasty using poly-L-D-lactic acid implant (RegJoint) interposition to fill the space left by resecting affected joint surfaces.
  Arms: Poly-L-D-lactic acid implant (RegJoint) interposition arthroplasty

SUMMARY:
This is a late (about 15 years) follow-up study of a randomized prospective clinical study originally conducted as a collaboration of the Rheumatism Foundation Hospital, Heinola, Finland and Päijät-Häme Central Hospital, Lahti Finland.

For the original study thirty-five patients with symptomatic end-stage inflammatory arthritis of the trapeziometacarpal joint were recruited. All patients signed written informed consent and were randomised to undergo surgery using either tendon interposition or poly-L-D-lactic acid implant interposition arthroplasty of said joint. The study was approved by the Päijät-Häme hospital district ethics committee.

Results of up to two years of follow-up have been published previously (DOI: 10.3109/2000656X.2012.669202).

For the current study all patients included in the final data analysis of the original study are to be contacted for a late follow-up using the same metrics used in the original study (hand pain and hand function rated on a visual analogue scale, hand strenght measurements, hand range of motion measurements, hand dexterity tests and tests simulating hand function in activities of daily living). Additionally outcomes will be assessed using the Patient Rated Wrist/Hand Evaluation and QuickDASH clinical outcome measurement scores.

Collected follow-up data will be statistically analyzed and a summary will be published in a peer-reviewed scientific journal.

ELIGIBILITY:
Inclusion Criteriria:

Patients of the study the results of which are reported in the following article: DOI: 10.3109/2000656X.2012.669202

Inclusion criteria for the original study:

* Symptomatic end- stage inflammatory arthritis of the trapeziometacarpal joint
* Trapeziometacarpal arthroplasty at Rheumatism Foundation Hospital, Heinola between january 2004 and december 2005
* Signed written informed consent

Exclusion criteria for the original study:

-age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Hand pain | Approximately 15 years from enrollment
  Pain of the studied / operated hand using a 0-100mm visual analogue scale where 0mm denotes no pain at all and 100mm denotes worst pain imaginable.
Hand function | Approximately 15 years from enrollment
  Function of the studied / operated hand using a 0-100mm visual analogue scale where 0mm denotes normal hand function and 100mm denotes the hand not functioning at all.
Hand grip strength | Approximately 15 years from enrollment
  Power grip strength (in kg) measured using a jamar hand dynamometer. Key pinch and tip pinch strength (in kg) mearured using a mechanical pinch gauge.
QuickDASH score | The previous week before approximately 15 years from enrollment
  The Disabilities of the Arm, Shoulder, and Hand (DASH) is a clinical outcome measure questionnaire consisting of thirty questions and has been validated several times. The QuickDASH score includes eleven of those questions and has been validated as well. Both scores are used to evaluate upper limb function and symptoms during the previous week.
Hand range of motion | Approximately 15 years from enrollment
  Active range of motion for following joints / parts of the hand: trapeziometacarpal joint radial abduction, thumb metacarpophalangeal joint extension and flexion, thumb interphalangeal joint extension and flexion.
Box and block dexterity test | Approximately 15 years from enrollment
  The Box and block dexterity consists of a rectangular box with a central dividing wall. The box is set on a table in front of the patient in a lengthwise orientation with the dividing wall at the patients midline. At the beginning of the test all 150 wooden cubes each 2,5cm are placed in the compartment on the side of the hand being tested. The test performed by moving as many 2,5cm wooden cubes one by one by hand from one box to another within 60 seconds as possible. Before the actual test the patient practices performing the test for 15 seconds with each hand,
Simulated activities of daily living tests | Approximately 15 years from enrollment
  Decanting water from a jug gripping the jug by its handle into a glass / cup. Decanting water from a glass / cup into jug gripping the glass with a palm grip. Cutting medical putty disc with knife and fork simulating cutting food on a plate.
  Picking up a wooden bead approximately 1cm in diameter using a pinch grip. The test is repeated four times for each hand so that the patient always uses their thumb but the opposing finger is different each time.
  Grading for all tests: Normal grip / adapted grip / unable to perform.
Radiological results | Approximately 15 years from enrollment
  Trapeziometacarpal joint (sub)luxation, joint trapeziometacarpal joint space height and bone destruction adjacent to the trapeziometarcpal joint using posterior to anteriot as well as lateral plain radiographs.
Patient Rated Wrist/Hand Evaluation clinical outcome measure | The previous week before approximately 15 years from enrollment
  The Patient-Rated Wrist and Hand Evaluation questionnaire is a region specific, patient reported outcome measure that aims to evaluate pain and disability of the wrist and hand. In one question the patient is asked about their hand / wrist today, while in fifteen questions the patient is asked about their hand / wrist this week. The score has been validated multiple times.

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided
At present we have no plan to share IPD as local legislature and the study protocol do not allow us to do so. If other researchers were to ask us to share IPD, we would be happy to apply permission to do so from our institution.

REFERENCES:
- [Background] Tiihonen RP, Skytta ET, Kaarela K, Ikavalko M, Belt EA. Reconstruction of the trapeziometacarpal joint in inflammatory joint disease using interposition of autologous tendon or poly-L-D-lactic acid implants: a prospective clinical trial. J Plast Surg Hand Surg. 2012 Apr;46(2):113-9. doi: 10.3109/2000656X.2012.669202. PMID 22471260